CLINICAL TRIAL: NCT06807411
Title: Investigation of the Effectiveness of a Video-Based Exercise Program Targeting Upper Extremity Function in Individuals With Parkinson
Brief Title: Effectiveness of Video-Based Upper Extremity Exercise Program in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-2282
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease; Exercise; Exergame; Therapy
Keywords: parkinson; exergame; serious game; exercise; physiotherapy
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional exercise group (Active Comparator): Participants in the conventional exercise group will undergo 24 sessions over 8 weeks (3 days per week, 30-minute sessions).
  The program will include:
  Stretching, strengthening, balance, gait, and posture exercises for the trunk and extremities.
  Kyphosis prevention exercises, including pectoral stretching, back extensor strengthening, and trunk mobilization.
  Resistance training using sandbags, dumbbells, and elastic bands. Tandem walking, weight-shifting on a balance board, and Frenkel coordination exercises.
  Each exercise will be performed for 15 repetitions, while stretching exercises will follow a 20-second stretch and 20-second rest protocol. Progression will be customized based on the participant's condition.
  Interventions: Other: Conventional exercise
- Video game based exercise group (Experimental): Participants will be randomly assigned to either a conventional exercise group or a video-based game exercise group. All participants will receive conventional therapy for 8 weeks, 3 days per week, with 30-minute sessions (24 sessions in total). The video-based game exercise group will undergo the same conventional therapy, with an additional video game-based exercise program using the Becure Extremity ROM device under physiotherapist supervision. The program will include KinectPong, KinectBalloon, ArmRotate, and Uball games. Balance, joint position sense, ROM, functionality, and quality of life parameters will be assessed before and after treatment.
  Interventions: Other: Video game based exercise

INTERVENTIONS:
Other: Conventional exercise — Participants in the conventional exercise group will receive a total of 24 sessions of conventional therapy over 8 weeks (3 days per week, 30-minute sessions).
  Arms: Conventional exercise group
Other: Video game based exercise — The video-based game exercise group will undergo the same conventional therapy, with an additional video game-based exercise program using the Becure Extremity ROM device under physiotherapist supervision. The program will include KinectPong, KinectBalloon, ArmRotate, and Uball games. Balance, joint position sense, ROM, functionality, and quality of life parameters will be assessed before and after treatment.
  Arms: Video game based exercise group

SUMMARY:
Over the past decade, virtual reality (VR) has been widely recognized as a therapeutic tool that enables neurological patients to interact with simulated environments through multiple sensory channels. Various sensors can be used in VR systems, with Nintendo Wii and Microsoft Kinect being the most popular. Video game-based training, grounded in VR technology, has emerged as a valid, cost-effective, and easily integrated adjunct to conventional therapy in neurorehabilitation. Compared to traditional exercise methods, video game training offers advantages by allowing users to perform physical activities in a safe and controlled environment. However, some studies have reported limited effects, emphasizing the need for more high-quality research to establish the effectiveness of interactive video games in neurological rehabilitation.

This study aims to investigate the effects of a video-based game exercise program targeting the upper extremity in individuals with Parkinson's disease on joint range of motion, proprioception, functionality, postural instability due to kyphotic posture, and quality of life.

DETAILED DESCRIPTION:
Over the past decade, virtual reality (VR) has been widely recognized as a therapeutic tool that enables neurological patients to interact with simulated environments through multiple sensory channels. Various sensors, such as Nintendo Wii and Microsoft Kinect, are commonly used in VR systems. Video game-based training has emerged as a valid, cost-effective, and easily integrated adjunct to conventional therapy in neurorehabilitation, offering a safe and controlled environment for physical activity. However, some studies have reported limited effects, highlighting the need for further high-quality research to establish its effectiveness in neurological rehabilitation.

This study aims to evaluate the effects of a video-based game exercise program targeting the upper extremity in individuals with Parkinson's disease on joint range of motion (ROM), proprioception, functionality, postural instability due to kyphotic posture, and quality of life. Participants will be randomly assigned to either a conventional exercise group or a video-based game exercise group. All participants will receive conventional therapy for 8 weeks, 3 days per week, with 30-minute sessions (24 sessions in total). The video-based game exercise group will undergo the same conventional therapy, with an additional video game-based exercise program using the Becure Extremity ROM device under physiotherapist supervision. The program will include KinectPong, KinectBalloon, ArmRotate, and Uball games. Balance, joint position sense, ROM, functionality, and quality of life parameters will be assessed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 50-80 with idiopathic Parkinson's disease
* Hoehn and Yahr Scale Stage I to III
* Presence of kyphotic posture

Exclusion Criteria:

* Presence of any other neurological condition
* Any pathology affecting the movement system in addition to Parkinson's disease
* Visual abnormalities
* Cardiovascular conditions that may interfere with treatment
* Dyskinesia
* History of surgery for Parkinson's disease
* Inability to cooperate at a level required to play the games

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Balance | From enrollment to the end of treatment at 8 weeks
  The Becure Balance System will be used to assess participants' postural stability. During this measurement, the participant will be asked to place both feet on the Balance Board and maintain balance for 15 seconds. Throughout this period, the participant's sway movements will be recorded.
Joint position sense | From enrollment to the end of treatment at 8 weeks
  The Becure Extremity ROM device will be used to assess proprioception in participants at 30° and 60° shoulder flexion and abduction positions. Participants will first be asked to raise their shoulder to a specified angle, then replicate the same angle with their eyes closed. The angle values recorded with eyes open and closed will be compared, and the difference between the shoulder angles will be calculated.
Range of motion | From enrollment to the end of treatment at 8 weeks
  joint range of motion (ROM) will be assessed using the Becure Extremity ROM system. This system utilizes built-in cameras and sensors to detect reference points during extremity movements, allowing for an objective measurement of joint ROM. In the Becure Extremity ROM assessment, the participant will stand in front of the camera and perform the required movement. Shoulder joint ROM, including flexion, extension, abduction, internal rotation, and external rotation, will be measured in degrees using this system.
Functionality | From enrollment to the end of treatment at 8 weeks
  Participants' upper extremity functionality will be assessed using the DASH (Disabilities of the Arm, Shoulder, and Hand) Questionnaire. DASH is designed to measure physical disability and symptoms in individuals with upper extremity disorders (hand, wrist, elbow, and shoulder). It is a 30-item scale that evaluates difficulties in performing various physical activities requiring upper extremity function.

SECONDARY OUTCOMES:
Parkinson's Disease Questionnaire (PDQ-39) | From enrollment to the end of treatment at 8 weeks
  Participants' quality of life will be assessed using the **Parkinson's Disease Questionnaire (PDQ-39)**. The **PDQ-39** is a self-administered tool that demonstrates optimal psychometric properties and reflects the full spectrum of quality of life in individuals with Parkinson's disease. The questionnaire consists of **39 items**.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Menek, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No